CLINICAL TRIAL: NCT02076776
Title: Heart-Brain Retraining: Forced Aerobic Exercise for Stroke Rehabilitation
Brief Title: Heart-Brain Retraining for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Jay Alberts, Principle Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R03HD073566 (NIH)
Record Dates: First submitted 2014-02-24; First posted 2014-03-04 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: Stroke; Exercise; Rehabilitation; Neuroplasticity; Task Practice
MeSH Terms: conditions — Stroke; Motor Activity | interventions — N-myc downstream-regulated gene 1 protein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Repetitive Task Practice (RTP) (Active Comparator): This group focuses on RTP.
  Interventions: Behavioral: Repetitive Task Practice (RTP)
- Voluntary cycling + RTP (Experimental): This group involves one biking session and one RTP session three times per week for eight weeks.
  Interventions: Behavioral: Voluntary cycling + RTP
- Assisted cycling + RTP (Experimental): This group involves one biking session and one RTP session three times per week for eight weeks.
  Interventions: Behavioral: Assisted cycling + RTP

INTERVENTIONS:
Behavioral: Repetitive Task Practice (RTP) — This group will preform arm and hand therapy.
  Arms: Repetitive Task Practice (RTP)
Behavioral: Voluntary cycling + RTP — This group will preform arm and hand therapy and cycle on a bike.
  Arms: Voluntary cycling + RTP
Behavioral: Assisted cycling + RTP — This group will preform arm and hand therapy and cycle on a bike.
  Arms: Assisted cycling + RTP

SUMMARY:
The purpose of this study is to gain a better understanding of how different types of exercise can help people after a stroke. The investigators want to study if different types of exercise will improve the use of arm and hand function after a stroke.

DETAILED DESCRIPTION:
Stroke is the leading cause of disability in the United States with approximately 795,000 new or recurrent strokes per year. An estimated two thirds of patients post-stroke cannot incorporate the affected upper extremity (UE) into their activities of daily living. In addition, stroke survivors experience a 60% decrease in cardiovascular capacity, which contributed to disability and diminished quality of life. Developing rehabilitation techniques to optimize motor recovery while improving cardiovascular endurance would benefit the stroke population.

Animal studies using a forced exercise (FE) paradigm, in which the rodent is exercised on a motorized treadmill at a rate greater than its voluntary rate, indicate an endogenous increase in neurotrophic factors such as brain-derived neurotrophic factor (BDNF) and glial-derived neurotrophic factor (GDNF). These neurotrophic factors are thought to underlie neuroplasticity and motor learning. It is hypothesized that patients with stroke, due to decreased motor cortical output, cannot sustain high rates of voluntary exercise necessary to trigger the endogenous release of neurotrophic factors; therefore, forced-exercise is necessary to augment their voluntary efforts and will be superior to voluntary exercise in facilitating motor recovery. When coupled with repetitive task practice (RTP) of the UE, an effective form of UE rehabilitation, FE will prime the brain for neuroplasticity. We have developed a safe and effective method of delivering forced-exercise to Parkinson's disease (PD) patients (NIH R21HD056316). Clinical and imaging data with PD patients indicate forced-exercise, but not voluntary exercise, triggers a neurophysiologic response in the central nervous system resulting in global improvements in motor and non-motor functioning and increased cortical and subcortical activation. The aim of this project is to conduct a preliminary trial to compare the effects of forced to voluntary exercise when coupled with RTP in promoting the recovery of motor function in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Within 6-12 months of diagnosis of single ischemic or hemorrhagic stroke, confirmed with neuroimaging
* Fugl-Meyer Motor Score 19-55 in involved upper extremity
* Approval from patient's primary care physician
* Age between 18 and 85 years

Exclusion Criteria:

* Hospitalization for myocardial infarction, congestive heart failure, or heart surgery (CABG or valve replacement) within 3 months of study enrollment
* Serious cardiac arrhythmia
* Hypertrophic cardiomyopathy
* Severe aortic stenosis
* Cardiac pacemaker
* Pulmonary embolus
* Other medical or musculoskeletal contraindication to exercise
* Significant cognitive impairment (unable to follow 1-2 step commands) or major psychiatric disorder (major depression, generalized anxiety) that will cause difficulty in study participation
* Anti-spasticity injection (botox) in upper extremity within 3 months of study enrollment
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Alberts, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Linder SM, Davidson S, Rosenfeldt A, Lee J, Koop MM, Bethoux F, Alberts JL. Forced and Voluntary Aerobic Cycling Interventions Improve Walking Capacity in Individuals With Chronic Stroke. Arch Phys Med Rehabil. 2021 Jan;102(1):1-8. doi: 10.1016/j.apmr.2020.08.006. Epub 2020 Sep 9. PMID 32918907
- [Derived] Linder SM, Davidson S, Rosenfeldt A, Penko A, Lee J, Koop MM, Phelan D, Alberts JL. Predictors of Improved Aerobic Capacity in Individuals With Chronic Stroke Participating in Cycling Interventions. Arch Phys Med Rehabil. 2020 Apr;101(4):717-721. doi: 10.1016/j.apmr.2019.10.187. Epub 2019 Nov 25. PMID 31778659
- [Derived] Rosenfeldt AB, Linder SM, Davidson S, Clark C, Zimmerman NM, Lee JJ, Alberts JL. Combined Aerobic Exercise and Task Practice Improve Health-Related Quality of Life Poststroke: A Preliminary Analysis. Arch Phys Med Rehabil. 2019 May;100(5):923-930. doi: 10.1016/j.apmr.2018.11.011. Epub 2018 Dec 10. PMID 30543801
- [Derived] Linder SM, Rosenfeldt AB, Rasanow M, Alberts JL. Forced Aerobic Exercise Enhances Motor Recovery After Stroke: A Case Report. Am J Occup Ther. 2015 Jul-Aug;69(4):6904210010p1-8. doi: 10.5014/ajot.2015.015636. PMID 26114455

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant consented to the study, but had abnormal stress test results. This participant declined follow-up care and withdrew from the study before completing the baseline and randomization process.
Period: Overall Study
Arm/Group | Repetitive Task Practice (RTP) | Voluntary Cycling + RTP | Assisted Cycling + RTP
Started | 6 | 8 | 6
Completed | 5 | 6 | 6
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Repetitive Task Practice (RTP) | Voluntary Cycling + RTP | Assisted Cycling + RTP | Total
Number analyzed (Participants) | 6 | 8 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 6 | 16
  >=65 years | 1 | 3 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.67 (7.45) | 59.38 (15.57) | 44.83 (11.72) | 55.70 (13.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 4
  Male | 6 | 5 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 4 | 6 | 3 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 6 | 20
Wolf Motor Function Test [Mean (Standard Deviation); unit: units on a scale] — Upper extremity function test. Total Functional Ability Score is reported. Scores range from 0-75 and higher scores indicate better function.
  units on a scale | 45.17 (17.38) | 49.75 (20.25) | 59.83 (9.06) | 51.40 (16.97)
Fugl-Meyer Assessment [Mean (Standard Deviation); unit: units on a scale] — Upper extremity motor test. Total score is reported. Scores range from 0-66 and higher scores indicate less impairment.
  units on a scale | 26.83 (7.83) | 34.75 (13.58) | 36.17 (7.41) | 32.80 (10.72)
Stroke Impact Scale [Mean (Standard Deviation); unit: units on a scale] — Quality of life questionnaire. Normalized Hand Function score is reported. Scores range from 0-100, with higher values indicating better self-reported quality of life.
  units on a scale | 31.67 (35.73) | 34.38 (28.72) | 50.83 (32.00) | 38.50 (31.29)

OUTCOME MEASURES:

1. Primary Outcome: Wolf Motor Function Test (WMFT)
Description: This consists of 2 strength tasks and 15 timed tasks of both the affected UE and the unaffected UE. Total Functional Ability Score is reported, scores range from 0-75, with higher scores indicating a better outcome.
Time Frame: Baseline, End of Treatment (8 weeks); End of Treatment + 4 week (12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Repetitive Task Practice (RTP) | Voluntary Cycling + RTP | Assisted Cycling + RTP
Number analyzed (Participants) | 5 | 6 | 6
units on a scale
  Baseline | 45.17 (17.38) | 49.75 (20.25) | 59.83 (9.06)
  EOT | 49.80 (18.94) | 48.83 (18.10) | 68.67 (6.31)
  EOT+4 | 50.80 (21.35) | 50.33 (19.35) | 69.50 (5.61)

2. Secondary Outcome: The Fugl-Meyer Assessment (FMA)
Description: This is a 33 item assessment of post-stroke UE impairment. Total score is reported, scores range from 0-66, with higher scores indicating a better outcome.
Time Frame: Baseline, End of Treatment (8 weeks); End of Treatment + 4 week (12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Repetitive Task Practice (RTP) | Voluntary Cycling + RTP | Assisted Cycling + RTP
Number analyzed (Participants) | 5 | 6 | 6
units on a scale
  Baseline | 26.83 (7.83) | 34.75 (13.58) | 36.17 (7.41)
  EOT | 29.80 (11.97) | 35.33 (14.65) | 48.50 (6.75)
  EOT+4 | 33.40 (15.04) | 37.00 (17.56) | 51.17 (3.06)

3. Other Pre Specified Outcome: The Stroke Impact Scale (SIS)
Description: This is a self-reported questionnaire evaluating quality of life. Normalized Hand Function is reported, scores range from 0-100, with higher scores indicating a better outcome.
Time Frame: Baseline, End of Treatment (8 weeks); End of Treatment + 4 week (12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Repetitive Task Practice (RTP) | Voluntary Cycling + RTP | Assisted Cycling + RTP
Number analyzed (Participants) | 5 | 6 | 6
units on a scale
  Baseline | 31.67 (35.73) | 34.38 (28.72) | 50.83 (32.00)
  EOT | 35.00 (26.93) | 45.00 (41.95) | 68.33 (15.38)
  EOT+4 | 34.00 (22.75) | 51.67 (37.24) | 66.67 (22.73)

ADVERSE EVENTS:
Arm/Group | Repetitive Task Practice (RTP) | Voluntary Cycling + RTP | Assisted Cycling + RTP
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Repetitive Task Practice (RTP) (N=6) | Voluntary Cycling + RTP (N=8) | Assisted Cycling + RTP (N=6)
Recurrent stroke (General disorders) | 0 (0) | 1 (1) | 0 (0) — One participant had a fatal recurrent stroke approximately 36 hours after the intervention. Upon reviewing the subject's medical history and stress test, the Patient Safety Monitoring Board unanimously concluded it was not due to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes